CLINICAL TRIAL: NCT04427293
Title: BRE-03: Window of Opportunity Trial of Preoperative Lenvatinib Plus Pembrolizumab in Early-Stage Triple-Negative Breast Cancer (TNBC)
Brief Title: Preoperative Lenvatinib Plus Pembrolizumab in Early-Stage Triple-Negative Breast Cancer (TNBC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Oana Danciu, Principal Investigator, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0232
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-07

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — lenvatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label (Experimental): All participants will receive lenvatinib 12mg daily for 7 days and pembrolizumab 200 mg IV on day 1 prior to surgery
  Interventions: Drug: Lenvatinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib 12mg daily for 7 days prior to surgery
Drug: Pembrolizumab — Pembrolizumab 200 mg IV on day 1

SUMMARY:
This is single arm study of a window of opportunity in which participants with previously untreated triple negative breast cancers (TNBC) who are candidates for potentially curative surgery will receive lenvatinib 12 mg daily for 7 and pembrolizumab 200 mg IV on day 1 prior to surgery

DETAILED DESCRIPTION:
This is a single arm study of a window of opportunity study in which participants with previously untreated triple negative breast cancers (TNBC) who are candidates for potentially curative surgery will receive therapy prior to surgery, consisting of lenvatinib 12 mg daily for 7 days and pembrolizumab 200 mg IV on day 1. Subjects will either have curative surgery 7-10 days after last dose of lenvatinib, and post-operative adjuvant therapy as per institution guidelines or have a research core biopsy of the breast tumor 7-10 days after last dose of lenvatinib, and standard of care neoadjuvant chemotherapy +/_ immune checkpoint inhibitor therapy, then curative surgery, post-operative adjuvant therapy as per institution guidelines

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age at time of consent
2. Histologically confirmed invasive breast carcinoma documented by core needle biopsy or incisional biopsy (excisional biopsy is not allowed). AJCC 8th edition clinical stage T1b-T3/N0-N3/M0 by physical exam or radiologic studies
3. Must be candidates for curative surgical resection
4. Have an FFPE diagnostic core biopsy specimen available that is determined by the study pathologist to be adequate for planned analyses
5. Definitive surgical excision of the primary breast tumor (either partial mastectomy or total mastectomy) and ipsilateral axillary lymph node sampling (sentinel lymph node biopsy or axillary dissection) is planned following completion of preoperative chemotherapy.
6. Estrogen Receptor (ER)- and Progesterone Receptor (PR)-negative as determined by immunohistochemistry (IHC), and Human Epidermal Growth Factor Receptor (HER)2-negative (triple-negative) cancer of the breast

   Triple-negative tumors are defined as:
   * Less than or equal to 10% of tumor cells staining for ER and for PR by immunohistochemistry (IHC)
   * HER2-negative, as defined by ASCO/CAP guidelines55
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 within 30 days prior to study registration
8. Demonstrate adequate organ function as defined in the table below; all screening labs to be obtained within 30 days prior to registration Hematological Leukocytes ≥2,500/mm3 Platelet count ≥ 100,000/mm3 Absolute Neutrophil Count (ANC) ≥ 1,500/mm3 Hemoglobin (Hgb) ≥ 9.0 g/dL Renal Creatinine/Calculated creatinine clearance (CrCl) Cr < 1.5 x upper limit of normal (ULN) or CrCl ≥ 50 mL/min using the Cockcroft-Gault formula Hepatic Bilirubin Bilirubin ≤ 1.5 × ULN. Subjects with Gilbert's syndrome may have a bilirubin > 1.5 × ULN, if no evidence of biliary obstruction exists Aspartate aminotransferase (AST) ≤ 2.5 × ULN Alanine aminotransferase (ALT) ≤ 2.5 × ULN
9. No evidence of distant metastases (M0 as per AJCC staging guidelines)
10. Provided written informed consent and HIPAA authorization for release of personal health information, approved by an Institutional Review Board (IRB)
11. NOTE: HIPAA authorization may be included in the informed consent or obtained separately
12. Women of childbearing potential (WOCP) must not be pregnant or breast-feeding. A negative serum or urine pregnancy test is required within 14 days of study registration. If the urine test cannot be confirmed as negative, a serum pregnancy test will be required
13. Women of childbearing potential (WOCP) must be willing to use two effective methods of birth control such as an oral, implantable, injectable, or transdermal hormonal contraceptive, an intrauterine device (IUD), use of a double barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream), or total abstinence for the course of the study until 120 days after the last dose of study drug NOTE: Women are considered to be of childbearing potential unless they are postmenopausal (≥45 years of age and has not had menses for greater than 12 consecutive months or bilateral oophorectomy) or surgically sterile (bilateral tubal ligation or hysterectomy) or not heterosexually active for the duration of the study and at least 120 days after the last dose of study drug
14. As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study

Exclusion Criteria:

1. Active infection requiring systemic therapy
2. Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study)
3. Previous anti-cancer treatment (cytotoxic chemotherapy, immunotherapy, biologic therapy, radiotherapy directed towards the primary breast tumor and/or ipsilateral axillary lymph nodes or investigational agents) with therapeutic intent for the current breast cancer
4. Previous treatment with lenvatinib or any immune checkpoint inhibitor within the past 2 years
5. Treatment with any investigational drug within 14 days prior to registration or within 5 half-lives of the investigational product, whichever is longer
6. Major surgery within 14 days prior to registration or has not recovered from major side effects of a major surgery (tumor biopsy and placement of an indwelling venous access device are not considered major surgery)
7. Any prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of this investigational regimen, as determined by the treating Medical Oncologist.
8. Known history of AIDS (HIV testing is not mandatory). HIV-positive individuals on active HARRT therapy with virologic suppression (defined as an HIV-1 RNA level below the lower limit of detection of the assay used) within 90 days of study enrollment and a CD4 cell count >500 cells/mm3 on the most recent determination are eligible for the study
9. . Subjects with any of the following conditions:

   * History of abdominal fistula, gastrointestinal perforation, or intra- abdominal abscess within 28 days prior to registration
   * History of cerebrovascular accident (CVA) or transient ischemic attack within 6 months prior to registration
   * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 6 months prior to registration
   * Symptomatic congestive heart failure (New York Heart Association III-IV) or documented current left ventricular (LV) systolic dysfunction with left ventricular ejection fraction (LVEF) <50% on most recent assessment of LV function
   * Clinically significant cardiac ventricular arrhythmias (e.g. sustained ventricular tachycardia/ventricular fibrillation) or high-grade AV block (e.g. bifascicular block, Mobitz type II and third-degree AV block) unless a pacemaker is in place
   * Any concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate subject participation in the clinical study or compromise compliance with the protocol
10. Any condition that, in the opinion of the investigator, might jeopardize the safety of the patient or interfere with protocol compliance
11. Any mental or medical condition that prevents the patient from giving informed consent or participating in the trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 12 (Estimated)
Dates: Start 2020-07-09 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of preoperative anti-vascular endothelial growth factor receptor (VEGFR) therapy and immune checkpoint blockade on infiltration of CD8+ tumor infiltrating lymphocytes (TILs) (CD45RA-/CD8+/FoxP3-) in primary tumors from patients | 2 years
  Measuring the presence of a T-cell inflamed TME, characterized by infiltration of CD8+ TILs

SECONDARY OUTCOMES:
Evaluate clinical response to preoperative anti-VEGFR therapy and immune checkpoint blockade based on pathologic complete response and residual tumor burden in subjects receiving neoadjuvant chemotherapy and changes in the Ki-67 index in all patients. | At the point of surgery
  Reviewing pathology report
Evaluate treatment tolerability of preoperative anti-VEGFR therapy and immune checkpoint blockade assessed by failure to completed planned course of neoadjuvant chemo-immune therapy and surgery in patients with early-stage TNBC | 30 days post treatment
  Assessing for adverse events (e.g., infections) using the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5

OTHER OUTCOMES:
Evaluate quality of life in patients with early-stage TNBC treated with preoperative anti-VEGFR therapy and immune checkpoint blockade | 5 years
  Reviewing questionnaires European Organization for Research, and Treatment of Cancer (EORTC) QLQ-C30 administered at screening, first post-op visit and final visit

CONTACTS AND LOCATIONS:
Overall Officials: Oana Danciu, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois, Chicago, Illinois, United States